CLINICAL TRIAL: NCT03962556
Title: Distribution of Trigger Points in Patient Who Have Myofascial Pain Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Funda Bastürk, Research assistant in Oral and Maxillofacial surgery, Necmettin Erbakan University
Other Study IDs: NecmettinEU1
Record Dates: First submitted 2019-02-19; First posted 2019-05-24 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Myofascial Pain
Keywords: trigger point,myofacial pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Trigger Point
  Interventions: Other: bimanual palpation
- Trigger Point
  Interventions: Other: bimanual palpation

INTERVENTIONS:
Other: bimanual palpation — bimanual palpation....i..

SUMMARY:
Myofascial pain alone covers 45.3% of the diagnosis of TMJ. It is defined as palpation sensitivity and regional muscle pain. Clinically muscle pain connects to myofascial trigger points.These trigger points are hypersensitive points located in a tense band of the skeletal muscle, which can be described, causing provoked or spontaneous pain. They are divided into two as active and latent. Those who cause spontaneous pain are active, and those who provoke pain are considered latent.Spasm in the chewing muscles with myofascial pain reduces the patient's pain threshold and quality of life.

Therefore, patients with spasm and TMJ pain in the masticatory muscles should be examined for head and neck muscles, the presence of myofascial trigger points should be determined and the head and neck muscles should be included in physical therapy.

The aim of this study was to determine the presence of myofascial trigger points in patients presenting with pain in the masticatory muscles and TMJ region, and to determine the relationship between the presence of trigger point and the degree of pain.

ELIGIBILITY:
Inclusion Criteria:

* Will be conducted in volunteers who applied to our clinic with complaint of TMJ

Exclusion Criteria:

* Diagnosed rheumatoid diseases and fibromyalgia.
* Psychiatric drug users.
* Patients who use muscle relaxants.
* TME pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Will be conducted in volunteers who applied to our clinic with complaint of TMJ
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
masticatory and cervical muscles examination for determining trigger points | first day visit
  detecting the trigger point (yes or no), determining the number of trigger points and determining the region on the muscle
visual analog scale for pain (VAS) | first day visit
  scale to find pain amount , pain scores from 0 to 10 will be taken from patients and higher scores indicate worse pain,all of patient's mean pain score to be determined.

SECONDARY OUTCOMES:
prevalence of trigger points in facial pain disorder patients | 1 year
  to compare pain scores of patients with and without trigger point,the distribution of trigger points on the masticatory and cervical muscles

CONTACTS AND LOCATIONS:
Overall Officials: Kubilay Işık, Study Chair — Necmettin Erbakan University/Dentistry Faculty; Dilek Menziletoğlu, Study Director — Necmettin Erbakan University/Dentistry Faculty; Funda Basturk, Principal Investigator — Necmettin Erbakan University/Dentistry Faculty
Locations (1):
- Necmettin Erbakan University/Dentistry Faculty, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided